CLINICAL TRIAL: NCT02070614
Title: Association of CYP3A4 rs2242480 With Sufentanil Plasma Concentration and PCA Consumption
Status: Completed | Type: Observational
Sponsor: Xianwei Zhang (Other)
Responsible Party: Sponsor-Investigator, Xianwei Zhang, Clinical Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: CYP3A4 and sufentanil
Record Dates: First submitted 2014-02-23; First posted 2014-02-25 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Surgery; Individuality
Keywords: sufentanil; metabolism; cytochrome P450 3A4; gene polymorphism

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — The blood samples were drawn before anesthesia，30 min and 45min after anesthesia respectively，used for genotyping and plasma sufentanil concentration detection with high performance liquid chromatography-mass spectrometry (HPLC-MS).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- rs2242480 wild-type homozygote: *1/*1 Grouped by rs2242480 polymorphism genotyping
- rs2242480 mutant heterozygote: *1/*1G Grouped by rs2242480 polymorphism genotyping
- rs2242480 mutant homozygote: *1G/*1G Grouped by rs2242480 polymorphism genotyping

SUMMARY:
This study was designed for exploring the association of cytochrome P450 3A4 rs2242480 polymorphism with metabolism of sufentanil in Chinese patients receiving upper abdominal surgery，to provide evidence for genetic prediction of personalized medication.Methods:60 patients who prepared for elective upper abdominal surgery under general anesthesia were recruited into study. Liver enzyme inhibitor should be excluded in anesthesia. rs2242480 genotyping was carried out by direct sequencing. The blood samples were drawn before anesthesia，30 min and 45min after anesthesia respectively，used for plasma sufentanil concentration detection with high performance liquid chromatography-mass spectrometry (HPLC-MS). After surgery，the patients received patient-controlled intravenous sufentanil immediately. And postoperative pain at rest，sufentanil consumption，side effects and rescue analgesic requirements were recorded at the 6th，12th，24th hour. The plasma sufentanil concentration and PCA sufentanil consumption were analyzed to investigate the differences among rs2242480 three genotypes.

DETAILED DESCRIPTION:
The study consisted of healthy men and women between 18 to 65 years of age.

Participants were screened and stratified according to cytochrome P450 3A4 rs2242480 genotype:

* 1/*1 Grouped by rs2242480 polymorphism, wild-type homozygote
* 1/*1G Grouped by rs2242480 polymorphism,*1/*1G: mutant heterozygote
* 1G/*1G Grouped by rs2242480 polymorphism,*1G/*1G: mutant homozygote

ELIGIBILITY:
Inclusion Criteria:

* 1.American Society of Anesthesiologists (ASA) physical status I or II 2.age from 18 to 65 years old 3.BMI of 19～26kg/m2

Exclusion Criteria:

* 1.known history of chronic pain, psychiatric diseases, diabetes mellitus, severe cardiovascular diseases, kidney or liver diseases with poor hepatic function 2.alcohol or drug abuse (according to the criteria of Diagnostic and Statistical Manual of Mental Disorders-IV) 3.pregnancy or at lactation period 4.Patients who consumed drugs (1 week) or foods (3 days) known to inhibit or induce the expression of cytochrome P450 3A4 enzymes prior to surgery were also excluded. The following drugs or foods included but were not limited to erythromycin, clarithromycin, alcohol, chocolate, coffee, grapefruit juice, verapamil, rifampicin, HIV protease inhibitors, phenytoin,itraconazole, dexamethasone, phenobarbital, and carbamazepine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 Chinese male and female patients receiving elective upper abdominal surgery (liver, pancreatic, gallbladder) under general anesthesia
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
the correlation between rs2242480 polymorphism and sufentanil metabolism | 4 months
  according to rs2242480 genotype and plasma concentration of sufentanil

SECONDARY OUTCOMES:
Variation of plasma concentration of sufentanil | 4 months
  the single-dose sufentanil plasma concentration varies between participants, and the differences among 3 time-points is related with personal genotype.
relation between rs2242480 genotype and patient-controlled analgesia(PCA) consumption of sufentanil | 4 months
  according to postoperative PCA sufentanil consumption and rs2242480 genotype
relation between Visual Analogue Scale/Score(VAS) and rs2242480 | 4 months
  according to PCA VAS and rs2242480 genotype

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, MD, Study Director — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China